CLINICAL TRIAL: NCT04588922
Title: A Phase I/IIa, Open-Label Dose Escalation and Dose Expansion Study of Intravenous GFH009 Single Agent and in Combination With Venetoclax and Azacitidine in Patients With Relapsed/Refractory Hematologic Malignancies
Brief Title: Study of SLS009 (Formerly GFH009) a Potent Highly Selective CDK9 Inhibitor in Patients With Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sellas Life Sciences Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GFH009X2101
Record Dates: First submitted 2020-09-28; First posted 2020-10-19 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancies
Keywords: Acute Myeloid Leukemia,; AML; Lymphoma; Chronic Lymphocytic Lymphoma; CLL; Small Lymphocytic Lymphoma; SLL; relapsed; refractory; CDK9 inhibitor; GFH009; SLS009; venetoclax; azacitidine; ASXL1
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Intervention Model Description: Open Label, Multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1. Dose escalation in patients with r/r AML (Experimental): In the dose escalation part, the dose levels will be escalated following the Bayesian optimal interval (BOIN) design. China study sites only. (Completed).
  Interventions: Drug: SLS009
- Group 2. Dose escalation in patients with r/r CLL/SLL or lymphoma (Experimental): In the dose escalation part, the dose levels will be escalated following the Bayesian optimal interval (BOIN) design. China and US study sites. (Completed).
  Interventions: Drug: SLS009
- Group 3 Cohort 1. 45 mg QW in patients with r/r AML (Experimental): SLS009 (45 mg QW) in combination with venetoclax and azacitidine in patients with r/r AML who have relapsed on or are refractory to venetoclax-based regimens. US study sites only. (Cohort completed)
  Interventions: Drug: SLS009; Drug: venetoclax; Drug: azacitidine
- Group 3 Cohort 2. 60 mg QW in patients with r/r AML. (Experimental): SLS009 (60 mg QW) in combination with venetoclax and azacitidine in patients with r/r AML who have relapsed on or are refractory to venetoclax-based regimens. US study sites only. (Cohort completed).
  Interventions: Drug: SLS009; Drug: venetoclax; Drug: azacitidine
- Group 3 Cohort 3. 30 mg BIW in patients with r/r AML. (Experimental): SLS009 (30 mg BIW) in combination with venetoclax and azacitidine in patients with r/r AML who have relapsed on or are refractory to venetoclax-based regimens. US study sites only. (Cohort completed).
  Interventions: Drug: SLS009; Drug: venetoclax; Drug: azacitidine
- Group 3 Cohort 4. 30 mg BIW in patients with r/r AML with ASXL1 mutation. (Experimental): SLS009 (30 mg BIW) in combination with venetoclax and azacitidine in patients with r/r AML who have relapsed or are refractory to venetoclax-based regimens and with documented ASXL1 mutation.
  Interventions: Drug: SLS009; Drug: venetoclax; Drug: azacitidine
- Group 3 Cohort 5. 30 mg BIW in pts with r/rAML with other than ASXL1 mutations (Experimental): SLS009 (30 mg BIW) in combination with venetoclax and azacitidine in patients with r/r AML who have relapsed or are refractory to venetoclax-based regimens and with documented Defining somatic mutations, Cytogenetic abnormalities defining acute myeloid leukemia, myelodysplasia related, other than ASXL1 mutation per WHO 5th Edition classification.
  Interventions: Drug: SLS009; Drug: venetoclax; Drug: azacitidine

INTERVENTIONS:
Drug: SLS009 — Solution for injection
  Other Names: GFH009
Drug: venetoclax — Tablets
  Other Names: Venclexta
  Arms: Group 3 Cohort 1. 45 mg QW in patients with r/r AML; Group 3 Cohort 2. 60 mg QW in patients with r/r AML.; Group 3 Cohort 3. 30 mg BIW in patients with r/r AML.; Group 3 Cohort 4. 30 mg BIW in patients with r/r AML with ASXL1 mutation.; Group 3 Cohort 5. 30 mg BIW in pts with r/rAML with other than ASXL1 mutations
Drug: azacitidine — Solution for injection
  Other Names: Vidaza; azacytidine
  Arms: Group 3 Cohort 1. 45 mg QW in patients with r/r AML; Group 3 Cohort 2. 60 mg QW in patients with r/r AML.; Group 3 Cohort 3. 30 mg BIW in patients with r/r AML.; Group 3 Cohort 4. 30 mg BIW in patients with r/r AML with ASXL1 mutation.; Group 3 Cohort 5. 30 mg BIW in pts with r/rAML with other than ASXL1 mutations

SUMMARY:
SLS009 (formerly GFH009) is a potent and highly selective CDK9 inhibitor. In this study the safety, tolerability, and antitumor activity of single agent SLS009 are assessed in two dose escalation groups (Group 1 in patients with relapsed/refractory AML, Group 2 in patients with relapse/refractory lymphoma/CLL/SLL). The safety, tolerability, and antitumor activity of SLS009 in combination with venetoclax and azacitidine in patient with relapsed/refractory AML who have relapsed on or are refractory to venetoclax-based regimens are being assessed in five cohorts of the expansion Group 3.

DETAILED DESCRIPTION:
SLS009 is a potent and highly selective CDK9 inhibitor. This study is investigating the safety, tolerability, and antitumor activity of SLS009 in patients with hematologic malignancies in three groups (two dose escalation groups and one expansion group). The safety and efficacy of SLS009 as a single agent are assessed in Group 1 (patients with relapsed/refractory AML) and Group 2 (patients with relapsed/refractory lymphoma/CLL/SLL). The safety and efficacy of SLS009 in combination with venetoclax and azacitidine in patients with relapsed/refractory AML who have relapsed on or are refractory to venetoclax-based regimens are being assessed in five different cohorts in the expansion Group 3. The cohorts in Group 3 include three cohorts to assess different dose levels (Cohorts 1, 2, and 3), a cohort enrolling patients with r/r AML and ASXL1 mutations and a cohort enrolling patients with r/r AML with other myelodysplasia-related mutations other than ASXL1.

ELIGIBILITY:
Inclusion Criteria

1. Male or female ≥ 18 years. and pediatric patients ages 12-18 and ≥40 kg body mass
2. Patients with cytological or histologically confirmed relapsed or refractory hematologic malignancies (AML, CLL/SLL and lymphoma)

   * Lymphoma: At least one measurable or evaluable lesion as defined by the Lugano (2014) response criteria. Patients must have received at least 2 prior lines of systemic therapy.
   * AML (only for Group 3): Patients relapsed on or refractory to venetoclax containing regimens.

     * AML, Cohort 4 (ASXL1 mutations): AML patients relapsed on and/or refractory to therapies containing venetoclax combinations and with documented ASXL1 mutation.
     * AML, Cohort 5 (Other than ASXL1 Myelodysplasia related AML defining somatic mutations): AML patients relapsed on and/or refractory to therapies containing venetoclax combinations and with documented Defining somatic mutations, Cytogenetic abnormalities defining acute myeloid leukemia, myelodysplasia related, other than ASXL1 mutation per WHO 5th Edition classification (The 5th edition of the World Health Organization Classification of Hematolymphoid Tumors: Myeloid and Histiocytic/Dendritic Neoplasms). Mutations in Cohort 5 include: BCOR, EZH2, SF3B1, SRSF2, STAG2, U2AF1 and ZRSR2. If any of those mutations is present concurrently with ASXL1 mutation, patients will be enrolled in Cohort 4 (ASXL1 mutation) and only patients harboring the above listed mutations without concurrent ASXL1 mutation will be enrolled in Cohort 5 (Other than ASXL1 Myelodysplasia related AML defining somatic mutations).
3. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) except for patients with Gilbert's syndrome, who are included if total bilirubin is < 3 × ULN or if direct bilirubin is < 1.5 × ULN.

   • Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN. For those with hepatic metastases, AST and ALT ≤ 5 × ULN.
4. Measured or calculated (determined by the Cockcroft-Gault equation) serum creatinine clearance (CrCl) ≥ 60 mL/min (glomerular filtration rate can be an alternative to CrCl).) for adult patients or serum creatinine ≤ 1.5 x ULN; or if serum creatinine > 1.5 x ULN, then serum creatinine clearance (CrCl) ≥ 50 mL/min (estimated by Cockcroft-Gault formula or other appropriate formula) for pediatric patients. Whether the value is calculated by equation or measured directly can be based on institutional standard practice.
5. Amylase ≤1.5 × ULN
6. Electrolytes and uric acid level need to be stable judged by investigators for at least 3 days before the first dose of SLS009 (formerly GFH009) (Medical intervention is permitted).
7. For women of childbearing potential, must consent to use highly effective methods (ie, total abstinence, placement of an intrauterine device) of contraception during SLS009 (formerly GFH009) treatment and for an additional 90 days after the last administration of study drug, if enrolled in Groups 1 or 2, and 6 months if enrolled in Group 3. Men with a partner of childbearing potential, must consent to use two highly effective methods of contraception during SLS009 (formerly GFH009) treatment and for an additional 90 days after the last administration of study drug.

Exclusion Criteria

1. Patients with bulky disease (≥ 10 cm) who require cytoreductive therapy.
2. Symptomatic central nervous system metastases or primary lymphoma such as primary CNS lymphoma, leptomeningeal disease, or spinal cord compression. Patients with asymptomatic CNS metastases who are radiologically and neurologically stable ≥ 4 weeks following CNS-directed therapy and are on a stable or decreasing dose of corticosteroids are eligible for study entry.
3. Severe cardiovascular disease within 6 months of study entry, including any of the following:

   * Clinically significant heart disease such as congestive heart failure requiring treatment (NYHA class III or IV), LVEF < 50% as determined by MUGA scan or echocardiogram (ECHO), (if only with historical occasional low LVEF but without any symptoms or relevant medical history, and the LVEF at screening is > 50%, the subject is eligible), or clinically significant arrythmia.
   * History/evidence of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting).
   * Average QTcF ≥ 450 msec (males) or ≥ 470 msec (females) on screening ECG.
   * Moderate or above regurgitation on echocardiogram
   * Patients with prior treatment with cardiotoxic agents who have experienced drug induced cardiotoxicities during or after treatment, where cardiotoxic agents include but are not limited to: anthracyclines (doxorubicin, daunorubicin, epirubicin, idarubicin, mitoxantrone); trastuzumab and trastuzumab based ADCs; tyrosine kinase inhibitors (sunitinib, imatinib); alkylating agents (cyclophosphamide).
   * Patients with a baseline cardiac biomarker abnormality (CKMB/cTnI) will be excluded.
4. Patients with hypereosinophilic syndrome defined as eosinophil counts in peripheral blood of ≥1,500/µ.
5. Concurrent malignancy within 5 years (for AML patients, 2 years) prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer not requiring treatment, ductal carcinoma in situ of the breast, and superficial non-muscle invasive urothelial carcinoma (excluding T1 lesions and CIS).
6. Active hepatitis B or hepatitis C virus infection.
7. History of HIV infection or HIV positive at screening.
8. Concomitant medications that are strong CYP3A4 inhibitors and strong inducers within 7 days prior to the first dose. Avoid consumption of Seville orange (and juice), grapefruit or grapefruit juice, grapefruit hybrids, pomelos, star citrus fruits or St. John's wort within 7 days of first dose.
9. Medications that are known to prolong the QT interval that could not be stopped prior to study entry judged by investigator, except azole antifungal medications in AML patients.
10. Subjects with high risk of gastrointestinal hemorrhage, including but not limiting to: active ulcer with fecal occult blood test ≥++; history of haematemesis or melena within 2 months prior first dose.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability: Dose Limiting Toxicities (DLTs) | 21 to 28 days
  The incidence of DLTs
Safety and Tolerability: adverse events (AEs) | approximately 2 years
  The incidence and severity of all AEs
Efficacy: ORR | 2 years
  Overall response rate is the proportion of patients showing anti-leukemic activity in response to treatment

SECONDARY OUTCOMES:
PK parameter AUC0-t | approximately 3 months
  Area under the plasma concentration-time curve (from zero to the time of the last measurable concentration)
PK parameter AUC0-∞ | approximately 3 months
  Area under the plasma concentration-time curve (from zero to infinity)
Efficacy: DOR | 2 years
  Duration of response in patients
Efficacy: PFS | 2 years
  Progression-free survival
Efficacy:OS | 2 years
  Overall survival
PK parameter Cmax | approximately 3 months
  Maximum plasma concentration reached following administration of study drug
PK parameter Tmax | approximately 3 months
  Time for maximum plasma concentration reached following administration of study drug
PK parameter t½ | approximately 3 months
  Half-life of study drug
Efficacy: ORR | 2 years
  Overall response rate is the proportion of patients showing anti-leukemic activity in response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Cicic, MD, Study Chair — SELLAS Life Sciences Group, Inc.
Locations (21):
- United States (8):
  - O'Neal Comprehensive Cancer Center, University of Alabama, Birmingham, Alabama
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Clinical Research Alliance, Inc., Lake Success, New York
  - New York - Presbyterian Hospital, New York, New York
  - UNC School of Medicine, Division of Hematology, Chapel Hill, North Carolina
  - Bon Secours St. Francis Cancer Center, Greenville, South Carolina
  - Baylor Scott & White Health, Dallas, Texas
  - MD Anderson, Houston, Texas
- China (13):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality
  - Cancer prevention and treatment center of Sun Yat sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shandong
  - Blood disease hospital, Chinese Academy of Medical Science, Tianjin, Tianjin Municipality
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No